CLINICAL TRIAL: NCT05990257
Title: Combined Multiple Regional Anesthesia for Microwave Ablation of Liver Tumors
Brief Title: CMRA for US-guided-MWA of Liver Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lu Wang (Other)
Responsible Party: Sponsor-Investigator, Lu Wang, Attending physician, Sichuan Cancer Hospital and Research Institute
Organization: Sichuan Cancer Hospital and Research Institute (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CMRA123
Record Dates: First submitted 2023-08-06; First posted 2023-08-14 (Actual); Last update posted 2023-08-15 (Actual); Status verified 2023-08

CONDITIONS: Regional Anesthesia; Pain Control; Microwave Ablation; Liver Tumors
MeSH Terms: conditions — Agnosia; Carcinoma, Hepatocellular

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HHB+TAPB+and LA (Experimental): Group A: patients who received a HHB, TAPB, and LA
  Interventions: Procedure: HHB+TAPB+and LA
- HHB+LA (Experimental): Group B: patients who received HHB and LA
  Interventions: Procedure: HHB+LA
- TAPB+LA (Experimental): Group C: patients who received TAPB and LA
  Interventions: Procedure: TAPB+LA

INTERVENTIONS:
Procedure: HHB+TAPB+and LA — Hepatic Hilar Block (HHB), Transversus Abdominis Plane Block (TAPB), and Local Anesthesia (LA)
  Arms: HHB+TAPB+and LA
Procedure: HHB+LA — Hepatic Hilar Block (HHB) and Local Anesthesia (LA)
  Arms: HHB+LA
Procedure: TAPB+LA — Transversus Abdominis Plane Block (TAPB) and Local Anesthesia (LA)
  Arms: TAPB+LA

SUMMARY:
Patients with liver tumors who underwent US-guided-MWA of liver tumors were enrolled. These patients were allocated into three groups based on tumor size and number: A, B, and C. Prior to the ablation procedure, Group A patients received a combination of hepatic hilar block (HHB), Transversus abdominis plane block (TAPB), and local anesthesia (LA). Patients in Group B were administered HHB in conjunction with LA, while those in Group C received TAPB and LA. Evaluative parameters included the Numerical Rating Scale (NRS) scores, consumption of morphine, incidence of complications, and factors influencing perioperative pain.

DETAILED DESCRIPTION:
Patients with liver tumors who underwent US-guided-MWA of liver tumors were enrolled. These patients were allocated into three groups based on tumor size and number: A, B, and C. Prior to the ablation procedure, Group A patients received a combination of hepatic hilar block (HHB), Transversus abdominis plane block (TAPB), and local anesthesia (LA). Patients in Group B were administered HHB in conjunction with LA, while those in Group C received TAPB and LA.Pain levels were routinely assessed through the Numerical Rating Scale (NRS), with scores being recorded by the attending nurse every 15 minutes. The frequency of these assessments would be increased if the patient reported discomfort or if there were changes observed in vital signs. If a patient reported a pain level of ≥4 on the NRS scale, an intravenous dose of 10mg morphine was administered, provided that cardiopulmonary safety could be assured. The determination of cardiopulmonary safety was made by the interventional radiologist (M. L. with 20 years of experience). Following the ablation procedure, all patients were monitored for a period of 36 hours. During this period, several parameters were recorded at the time of the procedure and again at 4, 8-, 12-, 24-, and 36-hours post-procedure. These parameters included the NRS score, vital signs, any need for morphine, and the occurrence of any adverse events.

ELIGIBILITY:
Inclusion Criteria:

Primary hepatic carcinoma was considered if characterized by a solitary tumor (≤5cm in maximum diameter) or by the presence of multiple tumors (2-3 in number, each ≤3cm in maximum diameter). Importantly, these tumors were required to be devoid of vascular invasion, biliary intrusion, contiguous organ invasion, or any evidence of distant metastasis.

Another group included in the study were patients with hepatic metastases, limited to no more than 5 tumors each measuring ≤3cm in maximum diameter.

Furthermore, patients with hepatic hemangioma were also considered for inclusion. Specific criteria applied in these cases included tumors larger than 5cm in maximum diameter that showed considerable growth (imaging findings suggest that the diameter of the tumor has increased by more than 1cm) in the preceding two years and were associated with persistent hemangioma-related abdominal pain or discomfort. Alternatively, tumors measuring up to 5cm in maximum diameter, exhibiting a pronounced growth propensity and located at the first, second, or third hilar region in close proximity to the hilar bile duct, portal vein, hepatic artery, hepatic vein, or inferior vena cava were also considered. And all these patients cannot tolerate surgery due to other organ damage or do not want to undergo surgical treatment.

The ASA grade is II or III.

Exclusion Criteria:

Patients with severe underlying medical conditions that could potentially prevent them from tolerating the US-guided MWA procedure were ruled out.

Those with tumors invading blood vessels, bile ducts, adjacent organs, or presenting with extrahepatic metastasis were also excluded.

Further, any cases presenting with uncorrectable coagulation disorders, thrombocytopenia, or currently under administration of anticoagulant agents were deemed unfit for the study.

Finally, patients were excluded if a safe trajectory for executing US-guided MWA was not feasible.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2018-07-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
pain control | at the time of the procedure and again at 4, 8-, 12-, 24-, and 36-hours post-procedure
  NRS score was used to evaluate pain control

CONTACTS AND LOCATIONS:
Overall Officials: Man Lu, PHD, Study Director — Sichuan Cancer Hospital and Research Institute
Locations (1):
- Sichuan cancer hospital, Chengdu, Sichuan, China